CLINICAL TRIAL: NCT00280098
Title: Phase IV Study of Safety and Efficacy of Docetaxel in Combination With Prednisone in Advanced Hormone Refractory Prostate Cancer Treatment
Brief Title: Docetaxel in the Treatment of Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Zuzana MD Priborska, Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_4001
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

ARMS (1):
- single group (Experimental)
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — Docetaxel 75mg/m2/q3wx10 cycles with Prednisone 10mg/d/bid

SUMMARY:
Evaluation of safety and efficacy of docetaxel in the treatment of advanced hormone refractory prostate cancer under the conditions of daily practise.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter :

Inclusion Criteria:

* Patients with advanced prostate cancer, without previous chemotherapy, progressing on hormonal treatment, performance status 1 to 2

Exclusion Criteria:

* Other cytostatic treatment, other malignity, severe comorbidity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
PSA decline | after each docetaxel administration and after the end of treatment
pain response | after each docetaxel administration and after the end of treatment
side effects occurrence | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana MD Priborska, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Prague, Czechia